CLINICAL TRIAL: NCT06922305
Title: A Study on the Relative Bioavailability of HR19042 Capsules in Healthy Subjects
Brief Title: Relative Bioavailability Study of HR19042 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HR19042-103
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Primary IgA Nephropathy; Autoimmune Hepatitis
MeSH Terms: conditions — Glomerulonephritis, IGA; Hepatitis, Autoimmune | interventions — Budesonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: HR19042 Capsules Period 2: Tarpeyo® Period 3: Budenofalk®
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®
- Sequence 2 (Experimental): Period 1: Tarpeyo® Period 2: Budenofalk® Period 3: HR19042 Capsules
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®
- Sequence 3 (Experimental): Period 1: Budenofalk® Period 2: HR19042 Capsules Period 3: Tarpeyo®
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®
- Sequence 4 (Experimental): Period 1: Tarpeyo® Period 2: HR19042 Capsules Period 3: Budenofalk®
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®
- Sequence 5 (Experimental): Period 1: HR19042 Capsules Period 2: Budenofalk® Period 3: Tarpeyo®
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®
- Sequence 6 (Experimental): Period 1: Budenofalk® Period 2: Tarpeyo® Period 3: HR19042 Capsules
  Interventions: Drug: HR19042 Capsule, Tarpeyo®, Budenofalk®

INTERVENTIONS:
Drug: HR19042 Capsule, Tarpeyo®, Budenofalk® — In each period under fasting conditions, subjects received oral administration of either HR19042 Capsule 16 mg, Tarpeyo® 16 mg, or Budenofalk® 15 mg.

SUMMARY:
This is a single-center, randomized, open-label, three-period, dual Latin square crossover study.

Primary Objective：

1. To evaluate the oral relative bioavailability of HR19042 Capsules compared with budesonide delayed-release capsules (Tarpeyo®) and budesonide enteric-coated capsules (Budenofalk®).

   Secondary Objective
2. To assess safety following administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ages 18 to 45, inclusive, at the time of informed consent.
2. Female subjects weigh ≥ 45 kg, male subjects weigh ≥ 50 kg, and BMI between 19.0 and 28.0 kg/m2, inclusive, at screening.
3. Understands the study procedures in the informed consent form ICF and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject with any history of severe allergic or anaphylactic reactions to any allergen including drugs, or allergic disease diagnosed and treated by a physician.
2. Clinically significant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine or connective tissue diseases or disorders
3. Subject has positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), or treponema pallidum antibody.
4. History of any gastrointestinal surgery or cholecystectomy that could impact the PK of study drugs.
5. Participated in other clinical trials within 3 months before screening or plan to participate in other clinical trials during this study.
6. Blood loss or blood donation of more than 300 mL within 3 months before screening, or intended to donate blood during the trial.
7. Those who have been vaccinated with vaccines within 3 month before screening or who have an intention to vaccinate during the trial.
8. Difficulty in venous blood sampling or fear of needles/blood.
9. Difficulty in swallowing capsules, or inability to comply with the provided diet and study-related instructions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum plasma concentration. Blood samples will be collected. | From Day 1 up to Day 8
AUC0-t: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected. | From Day 1 up to Day 8
AUC0-∞: Area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected. | From Day 1 up to Day 8
Tmax: Observed time to reach Cmax. Blood samples will be collected. | From Day 1 up to Day 8

SECONDARY OUTCOMES:
Incidence of treatment emergent AEs (TEAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided